CLINICAL TRIAL: NCT03780660
Title: Diagnostic Accuracy of the Central Venous Pressure (CVP) Variation to Predict Fluid Responsiveness in Spontaneously Breathing Patients
Acronym: VPVC
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017_60; 2018-A01449-46 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-12-18; First posted 2018-12-19 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Breathing
Keywords: Volume expansion; fluid responsiveness; critically ill patient; spontaneously breathing patient; central venous pressure variation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Volume expansion (VE) is often administered in intensive care (ICU)-patient to improve arterial oxygen delivery. Such effect is secondary to an increase in stroke volume and cardiac output. However, cardiac output increase in response to VE (fluid responsiveness) only occurs when the heart is preload-dependant. Increasing evidence of the deleterious effects of inappropriate fluid administration encourages the development of variables predicting fluid responsiveness, but few have been validated in spontaneously breathing patients.

Central venous pressure (CVP) variation in spontaneously patients during standardized or unstandardized inspiratory maneuver may represent an easy tool to predict fluid responsiveness. The hypothesise is that inspiratory maneuver may increase CVP variation in fluid responsiveness patient whereas no or few variation may reflect fluid unresponsiveness.

ELIGIBILITY:
Inclusion Criteria

* Spontaneous breathing without mechanical assistance
* Central venous catheter (superior vena cava) and monitoring of central venous pressure
* Urinary catheter and monitoring of intra-abdominal pressure

Exclusion Criteria:

* Intolerance to ventilatory manœuvre including Severe basal dyspnea/Symptomatic heart failure (pulmonary edema)
* Contraindication to passive leg raising (intracranial hypertension)
* Passive leg raising unsuitable for measuring hemodynamic response : High grade aortic insufficiency/ Poor echogenicity unsuitable to measure the velocity-time /integral of aortic blood flow/ Pregnancy/Abdominal hypertension with abdominal compartment syndrome/ Lower leg amputation
* Necessity of urgent hemodynamic therapy (within 90 min)
* Modification of hemodynamic therapy during study protocol (vascular filling, increase catecholamine dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient hospitalized in one of intensive care unit of Roger Salengro university hospital CHU Lille
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
the area under the ROC curve of the "CVPV-st" parameter | an average 60 - 90 minute during the procedure
  Diagnostic accuracy of the CVPV during a standardized inspiratory maneuver (CVPV-st) to predict fluid responsiveness.

SECONDARY OUTCOMES:
the area under the ROC curve of the "CVPV-un" parameter | an average 60 - 90 minute during the procedure
  Diagnostic accuracy of the CVPV during an unstandardized inspiratory maneuver (CVPV-un) to predict fluid responsiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Preau, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHU, Lille, France

REFERENCES:
- [Result] Bourel C, Durand A, Ter Schiphorst B, Martin C, Onimus T, De Jonckheere J, Howsam M, Pierre A, Favory R, Preau S. RESPIRATION-RELATED VARIATIONS IN CENTRAL VENOUS PRESSURE AS PREDICTORS OF FLUID RESPONSIVENESS IN SPONTANEOUSLY BREATHING PATIENTS. Shock. 2023 Aug 1;60(2):190-198. doi: 10.1097/SHK.0000000000002164. Epub 2023 Jul 26. PMID 37548683